CLINICAL TRIAL: NCT06793761
Title: A Prospective, Multicenter, Randomized Controlled Phase II Study to Evaluate the Efficacy and Safety of Salvage Preoperative PD-1 Inhibitor Combined with Chemotherapy Neoadjuvant Therapy in Recurrent and Metastatic Laryngeal and Hypopharyngeal Squamous Cell Carcinoma
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of Salvage Preoperative PD-1 Inhibitor Combined with Chemotherapy Neoadjuvant Therapy in Recurrent and Metastatic LPSCC/HPSCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRENT-002
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — pembrolizumab; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1-Pembrolizumab group (no previous radiotherapy) (Experimental): Patients who had not received RT previously received 3 cycles of pembrolizumab + cisplatin + nab-paclitaxel, followed by SOC treatment
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Nab-paclitaxel
- Arm 2 - Control group (no previous radiotherapy) (No Intervention): Patients who had not received RT before received SOC treatment only
- Arm 3 - Pembrolizumab group (previously received radiotherapy) (Experimental): Patients who had received RT before received 3 cycles of pembrolizumab + cisplatin + nab-paclitaxel, followed by SOC treatment
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Nab-paclitaxel
- Arm 4 - Control group (previously received radiotherapy) (No Intervention): Patients who had received RT before received SOC treatment only

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg, IV, 3 cycles
  Arms: Arm 1-Pembrolizumab group (no previous radiotherapy); Arm 3 - Pembrolizumab group (previously received radiotherapy)
Drug: Cisplatin — cisplatin 75mg/m2, IV, 3 cycles
  Arms: Arm 1-Pembrolizumab group (no previous radiotherapy); Arm 3 - Pembrolizumab group (previously received radiotherapy)
Drug: Nab-paclitaxel — Nab-paclitaxel 260mg, IV, 3 cycles
  Arms: Arm 1-Pembrolizumab group (no previous radiotherapy); Arm 3 - Pembrolizumab group (previously received radiotherapy)

SUMMARY:
A prospective, multicenter, randomized controlled phase II study; Patients who met the inclusion criteria were divided into groups according to whether they had received radical radiotherapy or postoperative radiotherapy in the past. Group A was the group that had not received radiotherapy in the past, and Group B was the group that had received radiotherapy. Group A was randomly given 3 cycles of pembrolizumab + chemotherapy (see P22 for detailed chemotherapy regimen) in the experimental group at a 1:1 ratio, followed by surgery. After surgery, the patients were stratified according to whether there were high-risk factors. The high-risk group received concurrent chemoradiotherapy + pembrolizumab maintenance therapy (up to 15 cycles), and the low-risk group received radiotherapy + pembrolizumab maintenance therapy (up to 15 cycles). The control group underwent direct surgery and received concurrent chemoradiotherapy or radiotherapy after surgery. The total dose of radiotherapy was (high-risk group: 60-66Gy, 2Gy/time; low-risk group: 44-50 Gy, 2Gy/time) adjuvant therapy, and the radiotherapy time was within 2 months after surgery. Group B was randomly given 3 cycles of pembrolizumab + chemotherapy in the experimental group at a ratio of 1:1, followed by surgery and maintenance therapy with pembrolizumab after surgery (up to 15 cycles). The control group was given surgery directly, and observation/re-radiotherapy or chemoradiotherapy was chosen by the doctor after surgery. The total dose of radiotherapy was (56-60Gy, 2Gy/time), and the radiotherapy time was within 2 months after surgery. The enrolled patients must be closely monitored for adverse reactions to chemotherapy, and the time, grade, treatment measures, and outcomes must be recorded. All patients received an examination after the end of neoadjuvant therapy, an examination after surgery, and an examination at the 9th week after the first radiotherapy, and then reviewed every 3 months for 1 year; after 1 year, they were reviewed once every 6 months for 3 years; the recurrence and survival data of the patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically and/or cytologically diagnosed squamous cell carcinoma of the larynx and hypopharynx
* Patients with recurrence of primary lesions or second primary lesions after definitive treatment
* At least 6 months from the end of the last platinum-containing treatment
* Cisplatin-tolerant
* Age ≥ 18 years
* ECOG 0-1
* Measurable disease as defined by RECIST v1.1
* Normal organ function
* Female and male participants of reproductive potential must agree to use appropriate contraception throughout the study and for 180 days after the last study treatment
* Male participants must not donate sperm throughout the study and for 180 days after the last study treatment

Exclusion Criteria:

* T stage after relapse (rT) is T4b
* Presence of distant metastasis
* Received live vaccines within 30 days before enrollment
* Diagnosed with immunodeficiency or received systemic steroids or any other form of immunosuppressive therapy within 7 days before enrollment
* Have radiologically detectable (even if asymptomatic and/or previously treated) central nervous system metastases and/or carcinomatous meningitis;
* Have undergone surgery before starting the study or have not recovered adequately from toxicity or complications caused by the intervention;
* Have had allogeneic tissue/solid organ transplantation;
* Have severe hypersensitivity reactions (≥ grade 3) to PD-1 inhibitors and chemotherapy or any of its adjuvants, radiotherapy;
* Have active autoimmune disease and require systemic treatment in the past 2 years;
* Have a history of (non-infectious) pneumonia requiring steroid treatment;
* Have a history of human immunodeficiency virus (HIV) infection;
* Any medical history, treatment, or laboratory abnormality that could confound the study results, interfere with the participant's participation throughout the study, or be detrimental to the participant's best interests;
* A known history of psychiatric or substance abuse disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate (2y-PFS rate) | 2 year
  To evaluate the 2y-PFS rate of neoadjuvant PD-1 inhibitors combined with chemotherapy in Arm 1 and Arm 3; PFS was defined as the time from patient enrollment to the occurrence of the following events (local progression/recurrence or distant metastasis (including neoadjuvant stage) assessed by imaging or biopsy, death from any cause)

SECONDARY OUTCOMES:
Pathological complete response rate (pCR rate) | 3 months
  To evaluate the pCR rate of neoadjuvant PD-1 inhibitors combined with chemotherapy in Arm 1 and Arm 3; pCR was defined as the absence of residual invasive squamous cell carcinoma cells in the resected primary tumor specimen and lymph nodes
Objective response rate (ORR) | 6 months
  To evaluate the ORR of neoadjuvant therapy with PD-1 inhibitors plus chemotherapy in Arm 1 and Arm 3; ORR is defined as The proportion of patients whose tumor volume shrinks to a pre-specified value and can be maintained for a certain period of time. It includes the proportion of patients with complete remission (CR) and partial remission (PR) to the total number of evaluable cases.
3-year overall survival rate (3y-OS rate) | 3 years
  To evaluate the 3y-OS rate of neoadjuvant PD-1 inhibitors plus chemotherapy in Arm 1 and Arm 3 in the overall population; OS was defined as the time from randomization until death from any cause.
Incidence of Treatment-Emergent Adverse Events (TRAEs) of pembrolizumab combined with chemotherapy in neoadjuvant therapy | 3 years
  TRAEs include 5 levels, base on Common Terminology Criteria for Adverse Events (CTCAE) is widely accepted as the standard classification and severity grading scale for adverse events in cancer therapy, clinical trials and other oncology settings.

IPD SHARING:
Plan to Share IPD: No